CLINICAL TRIAL: NCT00993850
Title: A Psychological Intervention for Individuals Who Suffer From Sleep Disturbance and Bipolar Disorder
Brief Title: Sleep Disturbance and Bipolar Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Allison Harvey, Professor of Clinical Psychology, National Institute of Mental Health (NIMH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34MH080958 (NIH); R34MH080958 (NIH); DAHBR A2-AID
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2013-04

CONDITIONS: Bipolar Disorder; Dyssomnias
Keywords: Bipolar disorder; Insomnia; Sleep disturbance; Cognitive behavioral therapy
MeSH Terms: conditions — Bipolar Disorder; Dyssomnias; Sleep Initiation and Maintenance Disorders; Parasomnias | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bipolar disorder education (Other): Psychoeducation
  Interventions: Other: Bipolar education
- Cognitive behavioral therapy (Other): Cognitive behavioral therapy for insomnia
  Interventions: Behavioral: Cognitive behavioral therapy for insomnia

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy for insomnia — Attending 6-10 treatment sessions in one of our interview rooms. The sessions will be offered on a weekly basis. Each session takes approximately 50 minutes.
  Arms: Cognitive behavioral therapy
Other: Bipolar education — Psychoeducation
  Arms: Bipolar disorder education

SUMMARY:
The study aims to evaluate a psychological intervention for individuals who suffer from sleep disturbance and bipolar disorder. We are hoping that this treatment will: (1) improve the quality of life of individuals with bipolar disorder who are suffering from sleep disturbance and (2) reduce the risk of, or help prevent, episodes.

ELIGIBILITY:
Inclusion Criteria:

Bipolar disorder patients with sleep disturbance

1. Meeting Diagnostic and Statistical Manual of Mental Disorders, 4th Text Revision (DSM-IV-TR; APA, 2000) diagnostic criteria for bipolar disorder type 1 (established with the SCID: Structured Clinical Interview for DSM-IV).
2. Being inter-episode throughout the experiment as defined by cutoffs widely used in previous research. On the basis that a drug-free group would likely be unfeasible and unrepresentative, participants will not be excluded on the basis of medications prescribed for bipolar disorder. Comorbidity will be allowed as long as bipolar disorder is the primary diagnosis. However, it is necessary to assess comorbidity for reporting purposes.
3. Participants who have a history of bipolar 1 or suicidal ideation must be under the care of a psychiatrist.
4. Experience distress related to significant sleep disturbance.

Exclusion Criteria:

1. Presence of an active and progressive physical illness (e.g., congestive heart failure, cancer, COPD) or neurological degenerative diseases (e.g., dementia, multiple sclerosis) directly related to the onset and course of insomnia;
2. Alcohol or drug abuse (except nicotine) within the past year
3. Active posttraumatic stress disorder
4. Evidence of sleep apnea, restless legs syndrome or periodic limb movements during sleep, or a circadian-based sleep disorder (e.g., delayed or advanced sleep phase syndrome)
5. Patients who pose a current suicidal risk or homicidal risk (assessed by treating psychiatrist) or who have made a suicide attempt within the past 6 months.
6. Pharmacotherapy for sleep defined as the benzodiazepine and non-benzodiazepine hypnotics that operate via the GABA A receptor complex and are FDA approved for the treatment of insomnia, selective melatonin agonists, benzodiazepine anxiolytics and over the counter medications with proven efficacy such as melatonin or herbs such as St. Johns wort.
7. Use of certain medications known to alter sleep (e.g., steroids, theophylline, propranolol, antihistamines that cause drowsiness).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-10; Primary Completion 2012-04 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Improvements in sleep, emotional functioning and quality of life | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University of California at Berkeley, Berkeley, California, United States